CLINICAL TRIAL: NCT04703140
Title: Evaluation of the Performance of COVIDISC Rapid Test for Diagnosis of SARS-CoV-2
Brief Title: COVIDISC: Rapid Diagnostic Tests on Nasopharyngeal Swabs for the Detection of COVID-19
Acronym: COVIDISC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Non-significant intemedial analysis
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/09
Record Dates: First submitted 2020-11-30; First posted 2021-01-11 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nasopharyngeal swabs (Experimental): One patient will have 2 nasopharyngeal for PCR and COVIDISC
  Interventions: Diagnostic Test: Rapid Diagnostic Test vs PCR

INTERVENTIONS:
Diagnostic Test: Rapid Diagnostic Test vs PCR — 2 nasopharyngeal swabs taken for PCR and COVIDISC

SUMMARY:
The Covid-19 pandemic requires a reliable diagnosis of patients in order to take care of them in the best conditions and in the appropriate services. Moreover, the current diagnostic reference is reverse transcription by polymerase chain reaction (RT-PCR) on a nasopharyngeal sample taken by swab. This technique is expensive (54€) and its production time is several hours.

Alternative methods are in progress, including, rapid diagnostic tests. The MEMS microfluids and nanostructures (MMN) laboratory, in partnership with the Institut Chimie Biologie Innovation (CBI) (Paris, 75005), have developed a portable test "COVIDISC", low-cost (10 €), fast (1 hour), including extraction, elution and amplification in solid medium isothermal, reverse amplification loop mediated transcription (RT-LAMP).

The "lab" version has received an analytical validation on human nasopharyngeal samples with performance comparable to classic RT-PCR (sensitivity of 7 copies per μl, specificity 100%).

The objective of this study is to validate the in vitro diagnostic medical device, COVIDISC, with the standard nasopharyngeal RT-PCR test.

DETAILED DESCRIPTION:
All outpatients and hospitalized patients (intensive care unit, internal medicine service and emergency service) will be proposed to participate to the study after assessment of eligibility criteria by the investigator. The investigator will collect a written consent of the patient or from the support person or a familiar if, the patient is not in condition to consent. Patient's participation will be notified in his medical record.

After inclusion of patient, the nurse will collect general and clinical data and 2 nasopharyngeal swabs will be taken. One sample to test the prototype of the RT-LAMP and the second one to carry out the classic RT-PCR. The results will be collected and compared in a second step.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing nasopharyngeal SARS CoV2 RT-PCR testing

Exclusion Criteria:

* < 18 years old
* Having signed a written informed consent form,
* Affiliation to the social security system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Comparaison of the performance of the diagnostic performance (sensitivity, sensibility) of RT-LAMP test using the RT-PCR test as a reference. | Day 0
  Calculate sensitivity, Specificity, Positive predictive value, Negative predictive value, Positive and negative likelihood report COVIDISC fast, antigenic test compared to RT-PCR Covid-19 reference test conducted in the laboratory

SECONDARY OUTCOMES:
Compare the diagnostic performances of RT-LAMP to clinical diagnosis. | Day 0
  The result of RT-LAMP test versus clinical evaluation defined by the clinical symptoms of the patients at the time of nasopharyngeal swab.

CONTACTS AND LOCATIONS:
Overall Officials: ROSSI Benjamin, MD, Principal Investigator — Hopital Robert Ballanger; NGUYEN Lee, MD, Principal Investigator — CMC Ambroise Paré
Locations (1):
- CHI Robert Ballanger, Aulnay-sous-Bois, France

IPD SHARING:
Plan to Share IPD: No